CLINICAL TRIAL: NCT04491097
Title: Clinical Outcomes of CAD/CAM Single-Retainer Monolithic Zirconia Ceramic Resin-Bonded Fixed Dentures Bonded With Two Different Resin Cements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Kuraray Noritake Dental Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E14107
Record Dates: First submitted 2020-07-14; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Denture, Partial, Fixed, Resin-Bonded; Tooth Loss / Rehabilitation; Resin Cements
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Panavia V5 resin cement (Experimental): Resin cement with non-MDP monomer
  Interventions: Device: Panavia V5 resin cement
- Experimental: Panavia F2.0 resin cement (Active Comparator): Resin cement with MDP monomer
  Interventions: Device: Panavia F2.0 resin cement

INTERVENTIONS:
Device: Panavia V5 resin cement — Missing lateral incisor teeth will be restored by zirconia ceramic RBFDs and adhesively bonded with Panavia V5 resin cement.The preperation and restoration of the tooth will be done according to to the guidelines for ordinary prosthetic techniques.
  Arms: Experimental: Panavia V5 resin cement
Device: Panavia F2.0 resin cement — Missing lateral incisor teeth will be restored by zirconia ceramic RBFDs and adhesively bonded with Panavia F2.0 resin cement.The preperation and restoration of the tooth will be done according to to the guidelines for ordinary prosthetic techniques.
  Arms: Experimental: Panavia F2.0 resin cement

SUMMARY:
Congenitally missing tooth is one of the most common anomalies in human dentition. The treatment options of lateral incisor agenesis are closing the space with orthodontic treatment, implant treatment, conventional fixed dental prosthesis (FDPs) and resin-bonded fixed dentures (RBFDs). RBFDs are used frequently for single tooth absence in the anterior region due to their minimal invasive properties, high clinical success and patient satisfaction. With the development of new and stronger materials, RBFDs with metal framework have been replaced by glass ceramic, lithium disilicate, fiber-reinforced composite (FRC) and zirconia. The aim of this study is to evaluate the clinical performance of CAD/CAM single-retainer monolithic zirconia ceramic RBFDs which cemented with two different resin cements.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical performance of CAD/CAM single-retainer monolithic zirconia ceramic RBFDs which cemented with two different resin cements.

The project includes 20 patients. Most of the patients have been recruited from the Istanbul Medipol University Dental Clinics in Istanbul. The patients were selected from individuals who have unilateral or bilateral congenitally missing maxillary lateral teeth and wanted to be treated a restoration or undergoing orthodontic treatment.

After giving their consent to take part in the study no preparations were made on abutment teeth for RBFDs. Digital impressions were taken with an intraoral digital scanner. The RBFDs were designed using a CAD software, milled and presintered zirconia blocks (KatanaTM Zirconia HT, Kuraray Noritake Dental Inc, Tokyo, Japan). RBFD was adhesively bonded to abutment teeth with one of the two different resin cements (Panavia F2.0 or Panavia V5).

The control procedure is:

The restoration is evaluated according to presence of mobility or debonding and fracture at the connector area. Gingival harmony and periodontal tissues around the restorations were also examined. Mobility of the abutment tooth was checked in the clinical examination and alveolar bone was examined with periapical x-ray. The controls will take place after two weeks, one year, two years, three years and five years.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the study voluntarily
* Horizontal mobility of central incisors ≤1 mm
* Central incisors with healthy alveolar bone
* 1-1,5 mm overjet
* Having a good anterior guidance

Exclusion Criteria:

* Patients with gingivitis or periodontitis Poor oral hygiene Central incisors with endodontic treatment or periapical disease Central teeth with large fillings or loss of dental structure on the cementation surface Bad oral habits Patients with clinical symptoms of bruxism

Ages: 18 Years to 80 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Survival rate of zirconia ceramic RBFDs | 5 years
  The survival was evaluated as described in the studies of Chai et al. (1). They described the survival as "the period of time starting at the cementation of the restoration and ending when the restoration was shown to have irreparably failed". The fracture was evaluated according to the study of Heintze and Rousson (2). They made a classification for fracture of zirconia restorations. Three grades of fracture treatment were assigned to this classification:
  (1) Grade 1: Fracture surfaces were polished. (2) Grade 2: Fracture surfaces were repaired with resin-based composite. (3) Grade 3: Severe chipping fractures required replacement of affected prostheses.
  1. Chai J, Chu FC, Newsome PR, et al: Retrospective survival analysis of 3-unit fixed-fixed and 2-unit cantilevered fixed partial dentures. J Oral Rehabil 2005;32:759-765
  2. Heintze SD, Rousson V. Survival of zirconia- and metal-supported fixed dental prostheses: a systematic review. Int J Prosthodont 2010;23:493-502

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No